CLINICAL TRIAL: NCT05861206
Title: Efficacy of Green and White Tea Extract Mouthwashes in the Management of Plaque-induced Gingivitis: A Clinical and Biochemical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yağmur Saraç Gül (Other)
Collaborators: Recep Tayyip Erdogan University (Other)
Responsible Party: Sponsor-Investigator, Yağmur Saraç Gül, one of principal investigator, Recep Tayyip Erdogan University
Organization: Recep Tayyip Erdogan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RecepTayyipErdoganU.1
Record Dates: First submitted 2023-03-26; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Gingivitis; Chronic; Oxidative Stress; Inflammation
Keywords: Green tea; White tea; Inflammation; Gingivitis; Oxidative stress
MeSH Terms: conditions — Gingivitis; Bronchiolitis Obliterans Syndrome; Inflammation | interventions — Tea

STUDY DESIGN:
Intervention Model Description: The inclusion criteria was as follows: presence of all primary teeth without a restoration, except the third molars; papillary bleeding index of 2 or 3 in at least 30% of papillae; no clinical attachment loss; being systemically healthy; and being normal weight according to body-mass index (BMI, 18,5-24,9 kg/m2). The exclusion criteria was as follows: usage of non steroidal anlgesics or antibiotics in last 6 months; usage of fixed or removable orthodontic appliance; presence of a intraoral soft tissue pathology; mouth breathing; smoking; a physical or mental disability that could prevent daily plaque control; and usage of any mouthwash in last 6 months.Chronic gingivitis patients aged 18-32 years whose mechanical plaque control was supported with different mouthwashes were randomly assigned into 4 groups of 28 people each: CHX-MW group (0.12% CHX, as a positive control group), EO-MW group (Listerine mouthrinse), GT-MW group (5% Green tea), and WT-MW group (5% White tea).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GT-MW group (5% Green tea), WT-MW group (5% White tea), EO-MW group (Listerine mouthrinse) (Active Comparator): Chronic gingivitis patients whose mechanical plaque control was supported with 5% Green tea. Each patient was instructed to use 15 mL of the mouthwash delivered to them for 60 seconds 30 minutes after brushing in the morning and evening for 4 weeks.
  Chronic gingivitis patients whose mechanical plaque control was supported with 5% White tea. Each patient was instructed to use 15 mL of the mouthwash delivered to them for 60 seconds 30 minutes after brushing in the morning and evening for 4 weeks.
  Chronic gingivitis patients whose mechanical plaque control was supported with Listerine mouthrinse. Each patient was instructed to use 15 mL of the mouthwash delivered to them for 60 seconds 30 minutes after brushing in the morning and evening for 4 weeks.
  Interventions: Other: GT-MW group (5% Green tea), WT-MW group (5% White tea),EO-MW group (Listerine mouthrinse)
- CHX-MW group (0.12% CHX, as a positive control group) (Active Comparator): Chronic gingivitis patients whose mechanical plaque control was supported with 0.12% CHX. Each patient was instructed to use 15 mL of the mouthwash delivered to them for 60 seconds 30 minutes after brushing in the morning and evening for 4 weeks.
  Interventions: Other: CHX-MW group (0.12% CHX, as a positive control group)

INTERVENTIONS:
Other: GT-MW group (5% Green tea), WT-MW group (5% White tea),EO-MW group (Listerine mouthrinse) — Subsequently, each patient was instructed to use 15 mL of the mouthwash (5% Green tea, 5% White tea or Listerine mouthrinse) delivered to them for 60 seconds 30 minutes after brushing in the morning and evening for a week. For the next 3 weeks, at the beginning of each week (8th, 15th and 22nd days), patients were invited to the clinic, oral hygiene instruction was repeated, and the mouthwashes to be used the following week were delivered to them.
  Arms: GT-MW group (5% Green tea), WT-MW group (5% White tea), EO-MW group (Listerine mouthrinse)
Other: CHX-MW group (0.12% CHX, as a positive control group) — Subsequently, each patient was instructed to use 15 mL of the mouthwash (0.12% CHX) delivered to them for 60 seconds 30 minutes after brushing in the morning and evening for a week. For the next 3 weeks, at the beginning of each week (8th, 15th and 22nd days), patients were invited to the clinic, oral hygiene instruction was repeated, and the mouthwashes to be used the following week were delivered to them.
  Arms: CHX-MW group (0.12% CHX, as a positive control group)

SUMMARY:
Background and objective: Tea is the second most consumed drink in the world after water. Gingivitis is among the most common infectious diseases. In this clinical study, Chlorhexidine Gluconate (CHX) was chosen as the positive control group and the clinical and biochemical efficacy of mouthwashes with green tea, white tea and essential oil (EO) as the active ingredients were aimed to be examined comprehensively.

Methods: 112 participants with gingivitis were randomly assigned to 4 different groups that different mouthwashes were used for 4 weeks. CHX-MW group (0.12% CHX, as a positive control group), EO-MW group (Listerine), GT-MW group (5% Green tea), and WT-MW group (5% White tea). The effects of the mouthwashes on plaque, inflammation, and dental staining were evaluated by indexed scores at the beginning and the end of the 4th week. In addition, markers related to gingival inflammation (IL-1beta, MMP-8) and oxidative stress (TOS, TAS, OSI (TOS/TAS)) were evaluated on samples from the gingival crevicular fluid.

DETAILED DESCRIPTION:
Chronic gingivitis patients aged 18-32 years whose mechanical plaque control was supported with different mouthwashes were randomly assigned into 4 groups of 28 people each: CHX-MW group (0.12% CHX, as a positive control group), EO-MW group (Listerine mouthrinse), GT-MW group (5% Green tea), and WT-MW group (5% White tea). The inclusion criteria was as follows: presence of all primary teeth without a restoration, except the third molars; papillary bleeding index of 2 or 3 in at least 30% of papillae; no clinical attachment loss; being systemically healthy; and being normal weight according to body-mass index (BMI, 18,5-24,9 kg/m2). The exclusion criteria was as follows: usage of non steroidal analgesics or antibiotics in last 6 months; usage of fixed or removable orthodontic appliance; presence of a intraoral soft tissue pathology; mouth breathing; smoking; a physical or mental disability that could prevent daily plaque control; and usage of any mouthwash in last 6 months.

All patients were given verbal and written motivational advice and modified bass brushing technique was taught on mouth models and in front of mirror. All patients were advised on brushes and toothpaste to use during the study period. Dental polishing was carried out if indicated. Subsequently, each patient was instructed to use 15 mL of the mouthwash delivered to them for 60 seconds 30 minutes after brushing in the morning and evening for a week. For the next 3 weeks, at the beginning of each week (8th, 15th and 22nd days), patients were invited to the clinic, oral hygiene instruction was repeated, and the mouthwashes to be used the following week were delivered to them.

Measurement of the clinical parameters and gingival crevicular fluid sample collection Clinical measurements ve gingival crevicular fluid (GCF) sample collection was carried out on each patient at the beginning of the study and at the end of the 4th week by a periodontist who was blinded about study group assignment.

Level of gingival inflammation was scored by mean of the following measurements: probing pocket depth (PPD) measured with a Williams type periodontal probe (Hu-Friedy, Chicago, Illionis, USA) on 6 different points (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual) around each tooth; plaque index (PI) ; and papillary bleeding index (PBI). In addition, the staining related to the mouthwash on the surface of the teeth and tongue was evaluated by gingival modification of the tooth staining index and tongue staining index in natural light environment. According to the tooth staining index, each tooth surface was divided into 4 separate regions and the staining intensity for each region was scored as; 0 = no staining, 1 = light staining (yellow), 2 = medium staining (brown), and 3 = intense staining (black). The staining index of the tongue was scored on the dorsal 2/3 front part of the tongue as; 0 = no staining, 1 = light staining (yellow), 2 = medium staining (brown), and 3 = intense staining (black). In the areas where two different colors were detected, the highest score was taken into account.

GCF samples were collected between 09.00 and 12.00, 24 hours after clinical periodontal parameters were recorded in order not to affect the current periodontal status of the patients. The samples were taken from a total of 4 teeth that each was with the most PPD in a seperate quadrant. Care was taken not to sample a tooth with caries or restoration on it and/or neighboring teeth. Samples were obtained by following steps: Supragingival plaque found in the region before sampling was removed by sterile curette. After isolating saliva with sterile cotton roll tampons, the region was dried with an air spray for 10 seconds without mechanical trauma. Paper strips in standard sizes (Periopaper; ProFlow, Inc., Amityville, NY, USA) was placed in 1mm depth in the sulcus and GCF was collected for 30 seconds (with the orifice technique). This step was repeated to collect a sufficient amount of samples. Strips contaminated with blood and saliva were not included in the study. The volume of GCF on each paper strip was measured by electronic impedance method (Periotron 8010, Oraflow Inc., NY, USA) in μl. 8 paper strips from the same patient were placed in a single ependorf tube with 250 μl of phosphate buffer (Phosphate Buffer Saline; PBS, pH = 7.4) and isolated from external environment by wrapping with parafilm (ISOLAB, Akron, Ohio, USA). The tubes were maintained at -80 oC (Thermo Fisher Scientific, Waltham, MA, USA) until the time of analysis.

Biochemical analysis IL-1beta and MMP-8 levels GCF IL-1beta and MMP-8 levels were determined in ng/ml using human-specific commercial ELISA kits (Elabscience Co, Ltd., Texas, USA).(Catalog no: H-0149 and H-1450, respectively) according to manufacturer instructions.

Measurement of TOS and TAS levels and Oxsidative Stres İndex (OSI) TOS and TAS levels were determined by automatic measurement method, using kits (Rel Assay Diagnostics, Gaziantep, Turkey) that were developed by Erel The results were expressed as μmol hydrogen peroxide (H2O2) equivalent/L and μmol Trolox equivalent/L. OSI was calculated by TOS/ TAS rate in percentage [(TOS (μmol H2O2 equivalents/L) / (TAS(μmol Trolox equivalent/L)].

Statistical analysis Statistical analyses were made with the help of IBM SPSS Statistics software (SPSS Inc., Chicago, USA) The normality of distribution was tested with Shapiro Wilk test. Inter group comparisons were made applying Kruskal Wallis, Mann Whitney U test, and Bonferroni correction. Wilcoxon test was applied for time-dependent changes within the groups. Differences in the level of p<0.05 were regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* all primary teeth without a restoration, except the third molars
* papillary bleeding index of 2 or 3 in at least 30% of papillae
* no clinical attachment loss; being systemically healthy
* being normal weight according to body-mass index

Exclusion Criteria:

* usage of non steroidal anlgesics or antibiotics in last 6 months
* usage of fixed or removable orthodontic appliance
* presence of a intraoral soft tissue pathology
* mouth breathing
* smoking
* a physical or mental disability that could prevent daily plaque control
* usage of any mouthwash in last 6 months

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Papillary bleeding index | changes of clinical findings from the beginning to 4th week
  A blunt periodontal probe was carefully inserted into the gingival sulcus at the base of the papilla on the mesial aspect, then moved coronally to the papilla tip. This was repeated on the distal aspect of the same papilla. Same procedure was followed on the lingual aspect of the papillas.The intensity of any bleeding thus provoked is recorded on a 0-4scale:
  Score 0:No bleeding Score I :A single discreet bleeding point appears Score 2: Several isolated bleeding points or a single fine line of blood appears Score 3:The interdental triangle fills with blood shortly after probing Score 4: Profuse bleeding occurs after probing; blood flows immediately into the marginal sulcus.
  Finally, scores are collected and calculate the arithmetic mean for the mouth score.
Plaque index | changes of clinical findings from the beginning to 4th week
  According to the tooth Plaque index, each tooth surface was divided into 6 separate regions and the plaque intensity for each region is scored as:
  0 = No plaque in the gingival area.
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
  Finally, scores are collected and calculate the arithmetic mean for the mouth score.
Probing pocket depth | changes of clinical findings from the beginning to 4th week
  Probing pocket depth (PPD) measured with a periodontal probe on 6 different points around each tooth. PPD is known as distance between gingival margin and the base of the pocket/sulcus. By using periodontal probe 6 different points are measured. Each scores of surfaces are collected and averaged for the mouth score for PPD.
Tooth staining index | changes of clinical findings from the beginning to 4th week
  According to the tooth staining index, each tooth surface was divided into 4 separate regions and the staining intensity for each region was scored as; 0 = no staining,
  1. = light staining (yellow),
  2. = medium staining (brown), and
  3. = intense staining (black). In the areas where two different colors were detected, the highest score was taken into account.
The staining index of the tongue | changes of clinical findings from the beginning to 4th week
  The staining index of the tongue was scored on the dorsal 2/3 front part of the tongue as; 0 = no staining,
  1. = light staining (yellow),
  2. = medium staining (brown), and
  3. = intense staining (black). In the areas where two different colors were detected, the highest score was taken into account.
Biochemical results:IL-1beta(ng/mL) | changes of biochemical findings from the beginning to 4th week
  IL-1beta(ng/mL), levels were determined in gingival crevicular fluid sample using human-specific commercial ELISA kits according to manufacturer instructions.
Biochemical results:MMP-8(ng/mL) | changes of biochemical findings from the beginning to 4th week
  MMP-8(ng/mL), levels were determined in gingival crevicular fluid sample using human-specific commercial ELISA kits according to manufacturer instructions.
Biochemical results:Total Oxidatif Status(μmol H2O2 Equiv./L) | changes of biochemical findings from the beginning to 4th week
  Total Oxidatif Status(TOS)(μmol H2O2 Equiv./L), levels were determined by automatic measurement method, using kits (Rel Assay Diagnostics, Gaziantep, Turkey) that were developed by Erel. The results were expressed as μmol hydrogen peroxide (H2O2) equivalent/L.
Biochemical results:Total Antioxidative Status(μmol Trolox. Equiv./L) | changes of biochemical findings from the beginning to 4th week
  Total Antioxidative Status(TAS)(μmol Trolox. Equiv./L) levels were determined by automatic measurement method, using kits (Rel Assay Diagnostics, Gaziantep, Turkey) that were developed by Erel. The results were expressed as μmol Trolox equivalent/L.
Biochemical results:Oxidative Stress Index[(μmol H2O2 Equiv./L)/(μmol Trolox. Equiv./L)] | changes of biochemical findings from the beginning to 4th week
  OSI was calculated by TOS/ TAS rate in percentage [(TOS (μmol H2O2 equivalents/L) / (TAS(μmol Trolox equivalent/L)].

CONTACTS AND LOCATIONS:
Locations (1):
- Yagmur Sarac Gul, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After publishing of this clinical trial, IPD will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: In a six month after the publication
Access Criteria: Study protocol, statistical analysis plan and clinical study repot will be shared.